CLINICAL TRIAL: NCT00178594
Title: Evaluation of Hemostasis in Bleeding and Thrombotic Disorders Using the Roteg Analyzer and the Thrombin Generation Assay
Brief Title: Evaluation of Hemostasis in Bleeding and Thrombotic Disorders
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Miguel Escobar, Professor - UTHealth McGovern Medical School, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-02-174
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Blood Coagulation Disorders, Inherited; Thrombotic Disorder
Keywords: Hereditary Bleeding disorder; Thrombotic Disorder
MeSH Terms: conditions — Blood Coagulation Disorders, Inherited; Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human whole blood and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this study will be to assess the coagulation system in-vitro in a variety of bleeding and clotting disorders using the ROTEG analyzer and the thrombin generation assay.

DETAILED DESCRIPTION:
This is an exploratory study involving blood coagulation assays in a select group of individuals receiving treatment for their congenital or acquired bleeding or clotting disorder at UTHealth Houston. The ROTEG is a newly developed coagulation analyzer which allows the continuous assessment of whole blood coagulation from the formation of the first fibrin fibers and activated platelets, to the formation of a three-dimensional whole blood clot until the eventual dissolution of the clot. This device will not be used as a diagnostic or procedure tool. No recommendations regarding interpretation of the results or implications for future treatment will be provided.

ELIGIBILITY:
Inclusion Criteria: patients with congenital or acquired bleeding or clotting disorders who have provided informed consent and/or assent

Exclusion Criteria: poor venous access

Ages: 1 Day to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with an acquired or congenital bleeding disorder or acquired thrombotic disorder receiving treatment for their condition at UTHealth Houston.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assess primary and secondary hemostasis in individuals with bleeding and clotting disorders | 24 hours
  Coagulation will be assessed by continuously recording clot firmness, thrombin generation, and platelet function

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Escobar, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The Univerisity of Texas Health Science Center at Houston, Houston, Texas
  - UT Physicians Women's Center-Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time